CLINICAL TRIAL: NCT04770324
Title: Monocentre, Non-Randomised Clinical Study Evaluating the Efficacy and Safety of 2 Supraflow® v1.3 Medical Devices in Glaucoma Surgery
Brief Title: Study of a Novel Interposition Supraciliary Implant in Patients With Open Angle Glaucoma (SAFARI 2)
Acronym: SAFARI 2
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: All original protocol assessments through M36 were completed. M48/60 were amendment additions to assess long-term efficacy. A new SV22 device was developed, and all subsequent studies used it. Amendments reflected interest in outcomes, not safety.
Sponsor: Ciliatech (Industry)
Collaborators: Clinchoice Inc (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAFARI 2
Record Dates: First submitted 2021-02-23; First posted 2021-02-25 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Glaucoma, Open-Angle
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interposition supraciliary implant (Experimental): Any patients corresponding to inclusion / exclusion criteria
  Interventions: Device: Interposition supraciliary implant

INTERVENTIONS:
Device: Interposition supraciliary implant — Surgical placement of 2 interposition supraciliary implant in the supraciliary space

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of implanting 2 novel interposition supraciliary implant as a stand-alone therapy for lowering intraocular pressure (IOP) in patients with primary open angle glaucoma (POAG) who have failed at least one class of topical medical therapy

DETAILED DESCRIPTION:
22 patients will be included in this 36 months interventional study.

All patients shall be indicated for glaucoma surgery alone (not combined with cataract), and will undergo incisional glaucoma therapy, including a novel simplified surgical technique allowing placement of 2 interposition supraciliary permanent devices.

Several patient data like IOP, visual capacity or associated pharmacological treatments will be recorded pre and post-operatively all along the follow-up.

Purpose is to ensure device safety, and verify IOP and associated pharmacological treatment reduction after surgery, and evolution along follow-up.

ELIGIBILITY:
Inclusion criteria:

Patient:

1. Patient ≥ 50 years old
2. Patient dated and signed the informed consent form to participate in the study at first visit

   Eye:
3. Phakic, pseudophakic or aphakic eye
4. Has medically treated open-angle glaucoma (schaffer grade 3 and 4)
5. The optimal medical treatment against glaucoma for this eye has failed i. Preoperative treatment ≥ 2 molecules with target IOP not reached despite medication, ii. or IOP ≥ 21 mmHg under treatment, iii. or patient not compliant with treatment, iv. or patient intolerant to treatment
6. Having undergone at most one filtration surgery (trabeculectomy, deep sclerectomy, viscocanalostomy) for more than 3 months.
7. Having the indication for glaucoma surgery alone

Exclusion criteria

Patient:

1. Patient with visual acuity of the contralateral eye greater than LogMar 0.3. If no problems are detected at three months post surgery on at least the first 10 patients included, the study monitoring committee may propose to relax this non-inclusion criterion by setting the visual acuity of the contralateral eye above LogMar 0.7
2. Patient with a known allergy to any of the constituents of the products used in this study
3. Patient already included in another study
4. A person protected by law (temporary or permanent guardianship) or not capable of discernment

   Eye
5. Presenting with inflammatory glaucoma
6. Presenting with congenital glaucoma
7. Presenting with major traumatic glaucoma or neovascular glaucoma or iridocorneal endothelial syndrome (ICE syndrome)
8. Having had a non-surgical operational treatment (ultrasound, cyclophotocoagulation, etc.)
9. Having had eye surgery (other than glaucoma) less than 6 months ago
10. Closed angle, grade 1 or 2 Schafer OAG
11. Pre-existing ocular or systemic pathology that may cause post operative complications such as:

    * Clinically significant inflammation such as uveitis
    * Eye infection
    * Anterior segment neovascular disease
12. Severe dry eye syndrome
13. Severe blepharitis
14. Retinopathy which can lead to neovascular complications in the anterior segment
15. Eye of axial length <20 mm
16. Eye with lens dislocation or subluxation

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-04-23 (Actual); Primary Completion 2024-07-26 (Actual); Study Completion 2024-07-26 (Actual)

PRIMARY OUTCOMES:
Assess post-op IOP reduction | 6, 12, 24, 26, 48, 60 months
  Proportion of Eyes With Intraocular Pressure (IOP) Reduction of ≥ 20%
Assess post-op IOP clinical success | 6, 12, 24, 26, 48, 60 months
  Proportion of Eyes With Intraocular Pressure (IOP) < 21 mmHg

SECONDARY OUTCOMES:
Evaluate implant and surgical procedure safety | up to 60 months
  To evaluate the safety of the implant and the surgical procedure: To describe of all adverse events (AEs) throughout the study
Compare clinical success rate | Up to 60 months
  To compare the clinical success rate at 6, 12, 24, 36, 48 and 60 months to that of the Supraflow study in Armenia
assess rate of patients with a reduction in post-op IOP with or without combined treatments | Up to 60 months
  To describe the rate of patients with at least a 20%, 25%, 30% and 40% reduction in postoperative IOP, with or without combined medical treatments, at each visit
assess rate of patients with IOP less than or equal to 18 mmHg and less than or equal to threshold | Up to 60 months
  To describe the rate of patients with a post-operative IOP ≤ 18 mm Hg; as well as for a threshold ≤ 16 mm Hg
assess the rate of patients with a reduction of IOP post-operatively | Up to 60 months
  To describe the rate of patients with a reduction of post-operative IOP of least 5 mmHg
assess the mean and median reduction in IOP | Up to 60 months
  To describe the mean and median reduction in IOP between the baseline and each subsequent assessment
assess the rate of patients without medical treatment for glaucoma | Up to 60 months
  To describe the rate of patients without medical treatment for glaucoma at each visit
average rate of IOP reduction | Up to 60 months
  describe the average rate of IOP reduction vs baseline
assess IOP stability | Up to 60 months
  To describe IOP stability over at each visit, without further eye surgery, and without the use of anti-glaucoma or adjunctive therapies such as goniopuncture or needling
assess the rate of patients with no filtering bleb | Up to 60 months
  To describe the rate of patients with no filtering bleb
Average number of adjunctive therapies and follow up visits | Up to 60 months
  To describe the average number of adjunctive therapies (needling, goniopuncture) and follow up visits (including those which were scheduled and which were not scheduled in the protocol)
Evaluate surgical procedure | Day 0, day of surgery
  To evaluate the surgical procedure (duration of operation, ease of implantation)
Assess patient satisfaction | Up to 60 months
  To describe patient satisfaction following surgery based on criteria of pain, discomfort and deterioration in visual acuity
Assess changes in quality of life | Up to 60 months
  To describe changes in quality of life (EQ5D)
Follow the progression of glaucoma and potential complications | Up to 60 months
  To describe the progression of the glaucoma at 6, 12, 24, 36, 48 and 60 months, and any complications

CONTACTS AND LOCATIONS:
Locations (1):
- Malayan Center, Yerevan, Armenia

IPD SHARING:
Plan to Share IPD: No